CLINICAL TRIAL: NCT03275974
Title: Glutamine PET Imaging of Colorectal Cancer
Brief Title: Glutamine PET Imaging Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: <75% participation
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-1083; NCI-2017-01543 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2017-08-30; First posted 2017-09-08 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-09

CONDITIONS: RAS Wild Type; Stage IV Colorectal Cancer; Stage IVA Colorectal Cancer; Stage IVB Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Magnetic Resonance Spectroscopy; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patients receive carbon C 11 Glutamine (11C-glutamine) IV and undergo PET imaging over 120 minutes. Beginning 2 hours to 7 days after 11C-glutamine PET, patients receive fluorine F 18 L-glutamate derivative BAY94-9392 (18F-FSPG) IV and also undergo PET imaging over 120 minutes. During each of the 11C-Glutamine and 18F-FSPG PET/CT scans, venous blood draws will be performed.
  Interventions: Biological: Carbon C 11 Glutamine; Biological: Fluorine F 18 L-glutamate Derivative BAY94-9392; Procedure: Positron Emission Tomography; Procedure: Blood Draw

INTERVENTIONS:
Biological: Carbon C 11 Glutamine — Given by IV
Biological: Fluorine F 18 L-glutamate Derivative BAY94-9392 — Given by IV
Procedure: Positron Emission Tomography — Undergo PET scan
Procedure: Blood Draw — Undergo venous blood draws

SUMMARY:
The clinical trial studies how well 11C-glutamine and 18F-FSPG positron emission tomography (PET) imaging works in detecting tumors in patients with metastatic colorectal cancer compared to standard imaging methods such as magnetic resonance imaging (MRI) or computed tomography (CT) scanning.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish and validate a 11C-glutamine (11C-Gln) and fluorine F 18 L-glutamate derivative BAY94-9392 (18F-FSPG) PET image guided gene signature to predict response to EGFR-targeted therapy in patients with advanced wild-type RAS colorectal cancer (CRC).

OUTLINE:

Patients receive 11C-glutamine intravenously (IV) and undergo PET imaging over 120 minutes. Beginning 2 hours to 7 days after 11C-glutamine PET, patients receive fluorine F 18 L-glutamate derivative BAY94-9392 IV and also undergo PET imaging over 120 minutes. During each of the 11C-Glutamine and 18F-FSPG PET/CT scans, venous blood draws will be performed.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age;
* Pathologically or cytologically confirmed diagnosis of metastatic (Stage IV) RAS wildtype CRC;
* Eligible for anti-EGFR monoclonal antibody (mAb) therapy as standard-of-care (SOC), either as a single agent or in combination with approved SOC therapies or investigational agents as part of IRB-approved clinical trials;
* Archived tissue from the CRC primary tumor in sufficient amounts to allow RNA-seq gene analysis; specimen from metastatic sites are not required but highly preferred;
* Documented results from (or scheduled to undergo) CT or MRI of the chest, abdomen and pelvis as a standard-of-care procedure within 28 days of baseline investigational 11C-Gln PET/CT and 18F-FSPG PET/CT;
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1;
* At least one lesion >2 cm in diameter and thus will be measurable according to PET Response Criteria in Solid Tumors (PERCIST) v1.0 to avoid PET partial volume effects;
* Ability to provide written informed consent in accordance with institutional policies.

Exclusion Criteria:

* Any other current or previous malignancy within the past 5 years
* Previous EGFR-directed therapy
* Body weight ≥ 400 pounds or body habitus or disability that will not permit the imaging protocol to be performed
* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2025-12-23 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
Pet imaging | Baseline prior to treatment with anti-EGFR mAb
  Assessed in terms of Standardized Uptake Values (SUVs)
Pharmacokinetic rate constants for 11C-Glutamine and 18F-FSPG | Baseline prior to treatment with anti-EGFR mAb
  The pharmacokinetic rate constants for 11C-Glutamine and 18F-FSPG will be determined using compartmental modeling of PET imaging data. Venous samples will be collected over the course of both 11C-Glutamine and 18F-FSPG scans for use in modeling.
Change in tumor size | Baseline prior to treatment with anti-EGFR mAb and every 8 weeks while on treatment (after every two (2) cycles of anti-EGFR mAb therapy (each cycle is 4 weeks)); through treatment completion, an average of 24 weeks (6 cycles)
  Change in tumor size will be derived from standard-of-care computed tomography (CT) or magnetic resonance imaging (MRI). The tumor size will be reported as either the long-axis diameter or as tumor volume.

SECONDARY OUTCOMES:
Gene expression | Prior to treatment with anti-EGFR mAb
  Gene expression will be determined using RNA-Seq of archived primary (and if available, metastatic) tissues.
Progression free survival | every 8 weeks while on treatment (after every two (2) cycles of anti-EGFR mAb therapy (each cycle is 4 weeks)); Up to 4 years after treatment
  Progression-free survival is defined as the time from start of therapy to disease progression by RECIST criteria or death for any reason.
Overall survival | Up to 4 years after treatment
  Overall survival is defined as the time from start of treatment to death for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Krebs, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2025-03-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT03275974/ICF_002.pdf